CLINICAL TRIAL: NCT06813378
Title: (Neuro)Cognitive Remediation for Adults With Operational Stress Injuries
Brief Title: (Neuro)Cognitive Remediation for Adults With OSIs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Abraham Rudnick, Clinical Director- Nova Scotia Operational Stress Injury Clinic, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 65194
Record Dates: First submitted 2025-01-31; First posted 2025-02-07 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: PTSD; Cognitive Impairment; Cognitive Dysfunction
Keywords: PTSD; Military; Veteran; Cognitive Remediation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will complete a minimum of 5 and a maximum of 17 one-on-one sessions (1-1.5 hrs in length) with an Occupational Therapist throughout the CR program. This program is designed to be tailored to a participant's individual needs, focusing on their specific cognitive impairments (hence the large range of potential sessions). During these sessions, participants will work with their clinician to learn compensatory strategies and restoration of cognition through a series of drill and practices to overcome their cognitive challenges.
  This study will use a mixed methods design incorporating both qualitative and quantitative research methods. Upon completion of the program, participants will be asked to complete a one-on-one interview with a researcher lasting approximately one hour. Additionally, participants will complete two psychometric questionnaires before beginning the cognitive remediation program and upon completion of the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- (Neuro)Cognitive Remediation (Experimental): Participants will undergo structured cognitive remediation program under the supervision of an Occupational Therapist. (Neuro)Cognitive Remediation will be achieved through teaching compensatory strategies, restoration of cognition through drill and practice and by utilizing regulative metacognitive strategies.
  Interventions: Behavioral: (Neuro)Cognitive Remediation

INTERVENTIONS:
Behavioral: (Neuro)Cognitive Remediation — (Neuro)Cognitive remediation is an intervention for people experiencing cognitive impairments that interfere with their daily functioning. Attention, memory, abstract reasoning, and processing speed are all examples of cognitive skills. By focusing on improving these underlying skills, the overall aim of cognitive remediation is to improve the client's daily satisfaction and success. Although cognitive remediation programs and strategies have been studied with other populations, it has not been sufficiently evaluated from a mental health trans-diagnostic perspective for military Veterans and police officers and retirees who this research will study.

SUMMARY:
(Neuro)Cognitive remediation (CR) is an intervention for people experiencing cognitive impairments that interfere with their daily functioning. Cognition refers to a person's ability to perceive, process, manipulate and respond to information. Attention, memory, abstract reasoning, and processing speed are all examples of cognitive skills. By focusing on improving these underlying skills, the overall aim of cognitive remediation is to improve the participant's daily satisfaction and success. CR can be achieved through teaching compensatory strategies, restoration of cognition through drill and practice and by utilizing regulative metacognitive strategies. Acquired skills and strategies are then 'bridged' or applied to daily functioning with the assistance of the clinician.

This pilot study intends to assess the impacts of a CR program on a population of Military Veterans, police officers, and retirees within the Nova Scotia Operational Stress Injury Clinic (NSOSIC). Researchers believe this program will improve cognitive functioning and that participants will perceive that the program was beneficial.

DETAILED DESCRIPTION:
CR is used in many client populations including acquired brain injury (ABI) , attention deficit hyperactivity disorder (ADHD) and post-traumatic stress disorder (PTSD) . Research has begun a more in-depth exploration into the relationship between psychological diagnoses and cognitive impairments. Difficulties in memory, attention, problem- solving ability, and processing speed have been linked to many mental health diagnoses which results in occupational dysfunction in the areas of daily routine, self-care, productivity, leisure, and relationships. Addressing these cognitive impairments with cognitive remediation can be an important step alongside other therapies in the recovery process.

Although CR programs and strategies have been studied with the populations referenced above, it has not been sufficiently evaluated from a mental health trans-diagnostic perspective for military Veterans and police officers and retirees. Additionally, the particular a combination of compensatory, restorative and regulative cognitive remediation used in the CR program for this research has not been published about for this clinical population that has cognitive impairments, but has been used with other populations of mental health service users .

Qualitative research methods will be the focus of this pilot study as they can provide a detailed understanding of the lived experiences of individuals using a relatively small sample size. Using qualitative research methodologies is also advantageous to answer the current research question as it allows participants to share experiences from their own point of view, rather than relying on the pre-suppositions of researchers, as would likely need to be done if trying to use quantitative research methods. Qualitative data will be obtained through individual semi-structured interviews with all participants of this study. These individual interviews will result in complete transcripts of conversations which can be thoroughly analyzed by researchers. This research will use an interpretive phenomenology framework for analysis, as will be described in the data analysis phase of this document.

Quantitative research methodologies will also be used within this pilot study. Four different psychometric measures will be completed by participants at the start and end of this study:

1. Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS)- a standardized assessment to screen for cognitive functioning which covers 5 domains: Immediate Memory, Visuospatial/Constructional, Language, Attention, and Delayed Memory.
2. World Health Organization Disability Assessment Schedule 2.0 (WHODAS)- a standardized assessment measuring health and disability across cultures which covers 6 domains: cognition, mobility, self-care, getting along, life activities, and participation.
3. Patient Health Questionnaire 9 Item (PHQ-9)- A 9-item screening tool used to assess the severity of depression-related symptoms.
4. Generalized Anxiety Disorder 7 Item (GAD-7)- a 7-item screening tool used to assess the severity of anxiety-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

Participants must be:

* Clients engaging in treatment at the Nova Scotia OSI Clinic who may benefit from the CR program.
* Be experiencing cognitive challenges which may be improved through the cognitive remediation program, as determined by the treating Occupational Therapist.

Exclusion Criteria:

Participants must not:

-Be accessing CR treatment modality through an Occupational Therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Participant Reported Qualitative Experience | From enrollment to the end of treatment- up to 17 weeks after enrollment.
  Qualitative data will be obtained through individual semi-structured interviews with all participants of this study. These individual interviews will result in complete transcripts of conversations which can be thoroughly analyzed by researchers. This research will use an interpretive phenomenology framework for analysis, as will be described in the data analysis phase of this document.

SECONDARY OUTCOMES:
1. Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS) | From enrollment to the end of treatment- up to 17 weeks after enrollment.
  A standardized assessment to screen for cognitive functioning which covers 5 domains: Immediate Memory, Visuospatial/Constructional, Language, Attention, and Delayed Memory. Total scale scores can range from 40-160, with lower scores indicating a worse outcome.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | From enrollment to the end of treatment- up to 17 weeks after enrollment.
  A standardized assessment measuring health and disability across cultures which covers 6 domains: cognition, mobility, self-care, getting along, life activities, and participation. Scores on this measure can range from 0-48, with higher scores representing a worse outcome.
Patient Health Questionnaire 9 Item (PHQ-9) | From enrollment to the end of treatment- up to 17 weeks after enrollment.
  A 9-item screening tool used to assess the severity of depression-related symptoms. Scores range from 0-27 with higher scores indicating higher levels of distress.
Generalized Anxiety Disorder 7 Item (GAD-7) | From enrollment to the end of treatment- up to 17 weeks after enrollment.
  A 7-item screening tool used to assess the severity of anxiety-related symptoms. Scores range from 0-21 with higher scores indicating higher levels of distress.
Montreal Cognitive Assessment | From enrollment to the end of treatment- up to 17 weeks after enrollment.
  a questionnaire administered by a trained clinician used to detect mild cognitive impairments with lower scores indicating cognitive impairment.

REFERENCES:
- [Background] Best MW, Bowie CR. A review of cognitive remediation approaches for schizophrenia: from top-down to bottom-up, brain training to psychotherapy. Expert Rev Neurother. 2017 Jul;17(7):713-723. doi: 10.1080/14737175.2017.1331128. Epub 2017 May 24. PMID 28511562
- [Background] Fonzo GA, Fine NB, Wright RN, Achituv M, Zaiko YV, Merin O, Shalev AY, Etkin A. Internet-delivered computerized cognitive & affective remediation training for the treatment of acute and chronic posttraumatic stress disorder: Two randomized clinical trials. J Psychiatr Res. 2019 Aug;115:82-89. doi: 10.1016/j.jpsychires.2019.05.007. Epub 2019 May 8. PMID 31125916
- [Background] McClure MM, Graff FS, Triebwasser J, Perez-Rodriguez MM, Rosell DR, Szeszko PR, Chu KW, New AS, Siever LJ, Hazlett EA. Neuroimaging predictors of response to cognitive remediation and social skills training: A pilot study in veterans with schizophrenia. Psychiatry Res Neuroimaging. 2019 Nov 30;293:110988. doi: 10.1016/j.pscychresns.2019.110988. Epub 2019 Oct 8. PMID 31655369
- [Background] Randolph C, Tierney MC, Mohr E, Chase TN. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity. J Clin Exp Neuropsychol. 1998 Jun;20(3):310-9. doi: 10.1076/jcen.20.3.310.823. PMID 9845158
- [Background] Stevenson CS, Whitmont S, Bornholt L, Livesey D, Stevenson RJ. A cognitive remediation programme for adults with Attention Deficit Hyperactivity Disorder. Aust N Z J Psychiatry. 2002 Oct;36(5):610-6. doi: 10.1046/j.1440-1614.2002.01052.x. PMID 12225443
- [Background] Twamley EW, Jak AJ, Delis DC, Bondi MW, Lohr JB. Cognitive Symptom Management and Rehabilitation Therapy (CogSMART) for veterans with traumatic brain injury: pilot randomized controlled trial. J Rehabil Res Dev. 2014;51(1):59-70. doi: 10.1682/JRRD.2013.01.0020. PMID 24805894
- [Background] Vanderploeg RD, Cooper DB, Curtiss G, Kennedy JE, Tate DF, Bowles AO. Predicting treatment response to cognitive rehabilitation in military service members with mild traumatic brain injury. Rehabil Psychol. 2018 May;63(2):194-204. doi: 10.1037/rep0000215. PMID 29878826